CLINICAL TRIAL: NCT06071715
Title: Cryoanalgesia to Treat Phantom Limb Pain Following a Trans-Femoral (Above-Knee) Amputation: A Randomized, Sham-Controlled Pilot Study
Brief Title: Cryoanalgesia to Treat Phantom Limb Pain Following Above-Knee Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRYO Pilot AboveKneeAmputation
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Amputation, Surgical; Amputation, Traumatic; Phantom Limb Pain; Phantom Pain Following Amputation of Lower Limb
MeSH Terms: conditions — Amputation, Traumatic; Phantom Limb | interventions — Cryosurgery

STUDY DESIGN:
Intervention Model Description: The primary endpoint at 1 month following the initial treatment will utilize a parallel group study design; however, an optional crossover is offered to subjects between 4-6 months following the initial treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All individuals will be masked to treatment with the exception of the anesthesiologist administering the procedure who will choose which probe to use: the functional or sham. Of note, this individual could not be masked to treatment since the cryoneurolysis ice ball is visualized on ultrasound; and, the practitioner would see a lack of ice ball formation for the sham probes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryoneurolysis first, then optional sham crossover treatment (Experimental): Initial treatment: Cryoneurolysis of the major nerves of the thigh in the residual limb: The cryoneurolysis device will be triggered using 1 cycle of 5.5-minute argon activation followed by a 30-60 second defrost with helium (Varian) or 2 cycles of 2-minute gas activation with an active probe separated by a 30-60 second defrost (Epimed). For active treatment, the gas will be deployed to the probe tip where a drop in temperature will result in cryoneurolysis.
  Optional sham crossover treatment: Sham cryoneurolysis of the major nerves of the thigh in the residual limb: The cryoneurolysis device will be triggered using 1 cycle of 5.5-minute argon activation followed by a 30-60 second defrost period with helium (Varian) or 2 cycles of 2-minute gas activation with a sham probe separated by a 30-60 second defrost (Epimed). However, for sham treatment, the gas is NOT deployed to the probe tip and therefore there is NO drop in temperature with NO resulting cryoneurolysis.
  Interventions: Device: ACTIVE cryoneurolysis; Device: SHAM cryoneurolysis
- Sham Comparator first, then optional cryoneurolysis treatment (Experimental): Initial treatment: Sham cryoneurolysis of the major nerves of the thigh in the residual limb: The cryoneurolysis device will be triggered using 1 cycle of 5.5-minute argon activation followed by a 30-60 second defrost period with helium (Varian) or 2 cycles of 2-minute gas activation with a sham probe separated by a 30-60 second defrost (Epimed). However, for sham treatment, the gas is NOT deployed to the probe tip and therefore there is NO drop in temperature with NO resulting cryoneurolysis.
  Optional active crossover treatment: Cryoneurolysis of the major nerves of the thigh in the residual limb: The cryoneurolysis device will be triggered using 1 cycle of 5.5-minute argon activation followed by a 30-60 second defrost period with helium (Varian) or 2 cycles of 2-minute gas activation with an active probe separated by a 30-60 second defrost (Epimed). For active treatment, the gas will be deployed to the probe tip where a drop in temperature will result in cryoneurolysis.
  Interventions: Device: ACTIVE cryoneurolysis; Device: SHAM cryoneurolysis

INTERVENTIONS:
Device: ACTIVE cryoneurolysis — Cryoneurolysis of the major nerves of the thigh (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 1 cycle of 5.5-minute argon activation followed by a 30-60 second defrost period with helium Initial treatment: Cryoneurolysis of the major nerves of the thigh (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 1 cycle of 5.5-minute argon activation followed by a 30-60 second defrost period with helium (Varian) or 2 cycles of 2-minute gas activation with an active probe separated by a 30-60 second defrost (Epimed). For active treatment, the gas will be deployed to the probe tip where a drop in temperature will result in cryoneurolysis.
  Other Names: cryoablation
Device: SHAM cryoneurolysis — SHAM cryoneurolysis of the major nerves of the thigh (or their distal counterparts) in the residual limb: The cryoneurolysis device will be triggered using 1 cycle of 5.5-minute argon activation followed by a 30-60 second defrost period with helium (Varian) or 2 cycles of 2-minute gas activation with a sham probe separated by a 30-60 second defrost (Epimed). However, for sham treatment, the gas is NOT deployed to the probe tip and therefore there is NO drop in temperature with NO resulting cryoneurolysis.
  Other Names: sham cryoablation

SUMMARY:
When a limb is severed, pain perceived in the part of the body that no longer exists often develops and is called "phantom limb" pain. Unfortunately, phantom pain goes away in only 16% of afflicted individuals, and there is currently no reliable definitive treatment. The exact reason that phantom limb pain occurs is unclear, but when a nerve is cut-as happens with an amputation-changes occur in the brain and spinal cord that actually increase with worsening phantom pain. These abnormal changes may often be corrected by putting local anesthetic-called a "nerve block"-on the injured nerve, effectively keeping any "bad signals" from reaching the brain with a simultaneous resolution of the phantom limb pain. However, when the nerve block resolves after a few hours, the phantom pain returns. But, this demonstrates that the brain abnormalities-and phantom pain-that occur with an amputation are not necessarily fixed, and may be dependent upon the "bad" signals being sent from the injured nerve(s), suggesting that a very long peripheral nerve block-lasting many months rather than hours-may permanently reverse the abnormal changes in the brain, and provide definitive relief from phantom pain. A prolonged nerve block lasting a few months may be provided by freezing the nerve using a process called "cryoneurolysis". The ultimate objective of the proposed research study is to determine if cryoanalgesia is an effective treatment for intractable post-amputation phantom limb pain. The proposed pilot study will include subjects with an existing above-knee amputation who experience intractable daily phantom limb pain. A single ultrasound-guided treatment of cryoneurolysis (or sham block-determined randomly like a flip of a coin) will be applied to the major nerves of the thigh. Although not required, each subject may return 4-6 months later for the alternative treatment (if the first treatment is sham, then the second treatment would be cryoneurolysis) so that all participants have the option of receiving the active treatment. Subjects will be followed for a total of 12 months with data collected by telephone.

DETAILED DESCRIPTION:
Subjects will be asked to make no changes to their analgesic regimen for at least 1 month prior to the cryoneurolysis procedure and continuing for 4 months until the measurement of the primary end point-for the duration of the study, all patients will be allowed to continue their pre-intervention analgesics. For individuals of childbearing potential, a sample of urine will be collected before any study interventions to confirm a non-pregnant state.

All subjects will have a peripheral intravenous catheter inserted, standard noninvasive monitors applied, and oxygen administered via a facemask or nasal cannula. Midazolam and/or fentanyl (IV) will be titrated for patient comfort.

Treatment group allocation (randomization). Participants will be allocated to one of two possible treatments groups:

1. Cryoneurolysis
2. Sham procedure (Control) Randomization lists will be created using computer-generated tables by the Investigational Pharmacy (UC San Diego) in a 1:1 ratio and block sizes of 2. Treatment group assignment will be conveyed to the investigators in the form of sealed, opaque envelopes only by the treating investigator. Therefore, all investigators and participants will be masked to treatment group assignment, with the only exception being the investigator and coordinator who perform the procedure (and will not have subsequent contact with the participant). This protocol will enable a randomized, observer- and participant-masked, sham/placebo-controlled study. It is impossible to mask the individual performing the cryoneurolysis procedure because the ice ball forming at the distal end of the probe-with active treatment-is clearly visible by ultrasound; and the lack of an ice ball for placebo participants is equally clear. It is essential to continuously visualize the probe and target nerve throughout the two freeze/thaw cycles to ensure the entire nerve diameter is adequately treated and remains relatively motionless. This cannot be achieved if the ultrasound is turned off during nitrous oxide administration to mask the provider; and the investigators prioritize patient safety over masking of the physician administering the intervention.

All participants will have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied (blood pressure cuff, pulse oximeter, 5-lead ECG), and oxygen administered via a nasal cannula or facemask. Midazolam and fentanyl (IV) will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues.

The cryoneurolysis sites will be cleansed with chlorhexidine gluconate and isopropyl alcohol. The nerves treated will include the femoral, sciatic, obturator, and lateral femoral cutaneous. Each nerve will be visualized using ultrasound, a skin wheal of local anesthetic will be raised inferior to the transducer to anesthetize the skin and then the track towards the target nerve. Participants randomized to active cryo will have 3-10 mL of ropivacaine 0.5% injected perineurally (20 mL maximum in total). The probe will then be inserted adjacent to the target nerve.

There are multiple types of cryoneurolysis machines cleared by the US FDA, all of which work on the same principle of a gas being passed through a small annulus, resulting in a dramatic pressure drop and accompanying temperature drop due to the Joule-Thomson effect. This study will utilize two different consoles: the Epimed International (Farmers Branch, TX) and Varian Medical Systems (Palo Alto, CA) machines. Which machine is used is determined by the size of the target nerve as judged by the administering physician: Epimed for smaller nerves (usually the obturator and lateral femoral cutaneous nerve) and Varian for larger (usually the sciatic and femoral nerves). There is no "accepted" diameter warranting the use of one vs the other, so this is left to the discretion of the physician.

Varian: This machine uses argon for the freeze cycle and helium to help decrease the thaw period duration. Sham probes are not available for this type of machine, and therefore an active probe will be used for all participants. For participants randomized to active treatment, the probe will be connected to the machine as usual, the argon (and helium) passed through the probe and then back into the machine, and finally vented out from the console. For participants randomized to sham treatment, the probe will simply not be connected to the back of the machine. For these participants the gas will simply be ejected directly from the console without ever having passed through the probe. The investigator administering the study intervention will attach the probe (active) or leave the tubing end close to the machine (sham).

Epimed: This machine uses nitrous oxide for the freeze cycle with a passive thaw (no gas flow). Cryoneurolysis probes are available that either (1) pass nitrous oxide to the distal end inducing freezing temperatures; or (2) vent the nitrous oxide at the proximal end of the probe so that no gas reaches the distal end, resulting in no temperature change. The latter is a sham procedure since without the temperature change, no ice ball forms and therefore the target nerve is not affected. Importantly, these probes are indistinguishable in appearance and will be differentiated only by an identifying stamp on the underside of the connector which is not visible during use. The investigator administering the study intervention will attach the appropriate probe to the cryoneurolysis device.

Varian: The cryoneurolysis machine (CryoCare, Varian Medical Systems, Palo Alto, California) uses argon for the freeze cycle and helium to help decrease the thaw period duration. The cryoneurolysis device will be triggered using 1 cycle of 5.5-minute argon activation followed by a 30-60 second helium defrost. The Varian machine provides its own timer so that the gas cycle timing is precise to the second. This may be repeated, as necessary, to ensure the entire cross-section of each nerve is fully treated.

Active Cryoneurolysis. For participants randomized to active treatment, the probe placed in the patient will be triggered and the argon (and helium) passed through the probe and then back into the machine, and finally vented out from the console. This will result in a freeze-thaw cycle.

Control. For participants randomized to sham treatment, the probe in the patient will simply not be activated; instead, a second probe that is not inserted in the patient will be triggered which will create the same visual and auditory cues as for the active participants retaining the masked feature. The investigator administering the study intervention will activate the correct probe depending on the treatment group assignment. Therefore, all investigators and participants will be masked to treatment group assignment, with the only exception being the unmasked investigator who performs the procedure (and will not have subsequent contact with the participant).

Epimed: The probe will be triggered using 2 cycles of 2-minute gas activation (active or sham) separated by a 30-60 second defrost. An observer (usually the research coordinator) will time the cycles and indicate to the investigator when the freeze and defrost periods have concluded to ensure adequate treatment duration.

It is impossible to mask the individual performing the cryoneurolysis procedure because the ice ball forming at the distal end of the probe-with active treatment-is clearly visible by ultrasound; and the lack of an ice ball for sham participants is equally clear. It is essential to continuously visualize the probe and target nerve throughout the freeze/thaw cycle(s) to ensure the entire nerve diameter is adequately treated and remains relatively motionless. This cannot be achieved if the ultrasound is turned off during nitrous oxide or argon administration to mask the provider; and the investigators prioritize patient safety over masking of the physician administering the intervention.

Prior to discharge, subjects will be provided with verbal and written instructions, the telephone and pager numbers of an investigator, and a copy of the Institutional Review Board-approved consent form. The approximate duration of this visit will total 4 hours, from the time the subject enters the treatment facility until the time the depart.

Optional crossover treatment. Four to six months following the initial treatment, subjects may return for an optional repeated intervention procedure ("crossover") with the alternative treatment (either active cryoneurolysis or sham/placebo), again in a double-masked fashion using the same protocol as described for the initial intervention. The crossover treatment is not required for study participation, as the primary analyses will include a parallel study design for the initial intervention evaluated prior to any crossover treatment. However, an optional crossover treatment will be offered to subjects for two reasons: (1) it will ensure that all subjects have access to the proposed treatment, regardless of the treatment participants are initially randomized to; and (2) it will permit intra-subject differences between treatments to be analyzed (e.g., assessing treatment-effect heterogeneity, or the variability of the causal effect across individuals, which will would not be available from the parallel-group portion of the study alone). These intra-subject differences will be secondary analyses, as there may be patient-selection bias regarding which subjects decide to have the crossover treatment (e.g., if the intervention is successful at greatly reducing phantom limb pain, then subjects receiving active cryoneurolysis during their initial treatment will be more likely to forgo the crossover treatment). This crossover will not affect the primary analyses, which will involve a parallel group study design and investigate the effects of cryoneurolysis within 4 months of the initial intervention. The approximate duration of a crossover visit will total 4 hours, from the time the subject enters the treatment facility until the time the depart. Following study completion, the results will be provided to all enrolled subjects using non-technical (i.e. "layperson") language, along with their treatment group assignment at the participants' request.

Following study completion, the results will be mailed electronically or by the United States Postal Service to all enrolled participants in written form using non-technical (e.g., "layperson") language.

Statistical analysis: Balance on baseline covariates will be assessed using absolute standardized difference (ASD); i.e., difference in means or proportions divided by the standard deviation. ASD > 0.1 will be considered to indicate imbalance, and these variables will be adjusted for in the statistical analyses. Analyses will be carried out using modified intention-to-treat; i.e., patients who received any study treatment will be analyzed according to the group participants were randomized to. Continuous, normally distributed data will be reported as mean ± standard deviation. Nonparametric continuous or categorical data will be reported as median [10th-90th percentiles] or percent, as appropriate. Comparisons of independent samples will be performed using Student's t-test for parametric continuous variables or Mann-Whitney U test for nonparametric or categorical variables. The Chi Square test and Fisher's Exact test will be used for differences in proportions, as appropriate. P<0.05 will be considered statistically significant for the primary and secondary outcomes with no correction for multiple comparisons. Results of comparisons in secondary outcomes will be interpreted as suggestive, requiring confirmation in a future trial before considering them as definitive.

Sample size determination: This is a pilot study to assist in powering a subsequent definitive trial and the investigators therefore use a convenience sample of 20 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients of at least 18 years of age
2. Trans-femoral traumatic or surgical amputation at least 12 weeks prior to enrollment distal to the hip (femoral head remaining)
3. Experiencing at least moderate phantom limb pain-defined as a 4 or higher on the Numeric Rating Scale (NRS; 0-10, 0= no pain; 10=worst imaginable pain)-at least daily for the previous 2 months
4. willing to avoid both changes to their analgesic regimen as well as elective surgical procedures from 1 month prior to and at least 4 months following the initial cryoneurolysis procedure.

Exclusion Criteria:

1. allergy to amide local anesthetics
2. pregnancy
3. incarceration
4. inability to communicate with the investigators
5. morbid obesity (body mass index > 40 kg/m2)
6. possessing any contraindication specific to cryoneurolysis such as a localized infection at the treatment site, cryoglobulinemia, cold urticaria and Reynaud's Syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Average pain intensity change from baseline 1 month post-intervention | Baseline and Month 1
  The "average" pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain. The primary outcome will be the change from baseline in average pain intensity as measured with the numeric rating scale 1 month following the initial intervention.

SECONDARY OUTCOMES:
Average Daily Phantom Pain intensity change from baseline | Post-intervention days 1, 7, and Months 2, 3, 4, and 12
  The "average" phantom pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Worst Daily Phantom Pain intensity change from baseline | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  The "worst" phantom pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Least Daily Phantom Pain intensity change from baseline | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  The "least" phantom pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Current Daily Phantom Pain intensity change from baseline | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  The "current" phantom pain level measured using the numeric rating scale at the time of the data collection phone call. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
CROSSOVER Average Daily Phantom Pain intensity change from baseline | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  The "average" phantom pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
CROSSOVER Worst Phantom Pain intensity change from baseline | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  The "worst" phantom pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
CROSSOVER Least Phantom Pain intensity change from baseline | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  The "least" phantom pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
CROSSOVER Current Phantom Pain intensity change from baseline | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  The "current" phantom pain level measured using the numeric rating scale at the time of the data collection phone call. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Average Daily Residual Limb Pain intensity change from baseline | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  The "average" residual limb pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Worst Daily Residual Limb Pain intensity change from baseline | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  The "worst" residual limb pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Least Daily Residual Limb Pain intensity change from baseline | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  The "least" residual limb pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Current Residual Limb Pain intensity change from baseline | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  The "current" residual limb pain level measured using the numeric rating scale at the time of the data collection call. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
CROSSOVER Average Daily Residual Pain intensity change from baseline | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  The "average" residual limb pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
CROSSOVER Worst Daily Residual Pain intensity change from baseline | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  The "worst" residual limb pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
CROSSOVER Least Daily Residual Pain intensity change from baseline | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  The "least" residual limb pain level measured using the numeric rating scale for the previous 24 hours. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
CROSSOVER Current Residual Pain intensity change from baseline | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  The "current" residual limb pain level measured using the numeric rating scale at the time of the data collection phone call. This is a 0-10 Likert scale measuring pain level with 0=no pain and 10=worst imaginable pain.
Patient Global Impression of Change, Initial intervention | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  This measure is a 7-point ordinal scale requiring the subject to rate the current severity of their global situation as it relates to phantom limb pain (as defined by each individual) compared to their baseline. This scale has the words "very much worse" to the left by the number one, and "very much improved" to the right, adjacent to the number seven. The words "no change" are in the middle of the scale above the number four.
CROSSOVER Patient Global Impression of Change | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  This measure is a 7-point ordinal scale requiring the subject to rate the current severity of their global situation as it relates to phantom limb pain (as defined by each individual) compared to their baseline. This scale has the words "very much worse" to the left by the number one, and "very much improved" to the right, adjacent to the number seven. The words "no change" are in the middle of the scale above the number four.
Brief Pain Inventory (interference sub scale), initial intervention | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  The Brief pain Inventory (short form) is an instrument specifically designed to assess pain and its impact on physical and emotional functioning. The brief Inventory is comprised of three domains: (1) pain, with four questions involving "worst", "average" and "current" pain levels using a 0-10 numeric rating scale;(2) percentage of relief provided by pain treatments with one question [reported score is the percentage divided by 10 and then subtracted from 10: 0=complete relief,10=no relief] and, (3) interference with 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference;10=complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. This outcome will include the interference subscale.
CROSSOVER Brief Pain Inventory (interference sub scale) | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  The Brief pain Inventory (short form) is an instrument specifically designed to assess pain and its impact on physical and emotional functioning. The brief Inventory is comprised of three domains: (1) pain, with four questions involving "worst", "average" and "current" pain levels using a 0-10 numeric rating scale;(2) percentage of relief provided by pain treatments with one question [reported score is the percentage divided by 10 and then subtracted from 10: 0=complete relief,10=no relief] and, (3) interference with 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference;10=complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. This outcome will include the interference subscale.
Phantom Limb Pain Frequency, initial intervention | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  Number of occurrences of phantom limb pain experienced in the previous 24 hours
Phantom Limb Pain Duration, initial intervention | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  Average duration of each phantom limb pain experienced in the previous 24 hours
Residual Limb Pain Frequency, initial intervention | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  Number of occurrences of residual limb pain experienced in the previous 24 hours
Residual Limb Pain Duration, initial intervention | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  Average duration of each residual limb pain experienced in the previous 24 hours
Non-painful phantom sensations Frequency, initial intervention | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  Number of occurrences of non-painful phantom sensations experienced in the previous 24 hours
Non-painful phantom sensations Duration, initial intervention | Post-intervention days 1, 7, and Months 1, 2, 3, 4, and 12
  Average duration of non-painful phantom sensations experienced in the previous 24 hours
Phantom Limb Pain Frequency, CROSSOVER intervention | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  Number of occurrences of phantom limb pain experienced in the previous 24 hours
Residual Limb Pain Frequency, CROSSOVER intervention | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  Number of occurrences of residual limb pain experienced in the previous 24 hours
Phantom Limb Pain Duration, CROSSOVER intervention | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  Average duration of each phantom limb pain experienced in the previous 24 hours
Residual Limb Pain Duration, CROSSOVER intervention | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  Average duration of each residual limb pain experienced in the previous 24 hours
Non-painful phantom sensations Frequency, CROSSOVER intervention | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  Number of occurrences of non-painful sensations experienced in the previous 24 hours
Non-painful phantom sensations Duration, CROSSOVER intervention | Following the CROSSOVER treatment on Days 1 and 7; Months 1, 2, 3, and 4
  Average duration of non-painful sensations experienced in the previous 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ilfeld, MD, MS, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gabriel RA, Finneran JJ 4th, Trescot AM, Ilfeld BM. Ultrasound-Guided Percutaneous Cryoneurolysis for Postoperative Analgesia After Limb Amputation: A Case Series. A A Pract. 2019 Apr 1;12(7):231-234. doi: 10.1213/XAA.0000000000000893. PMID 30234513
- [Background] Said ET, Marsh-Armstrong BP, Fischer SJ, Suresh PJ, Swisher MW, Trescot AM, Prologo JD, Abdullah B, Ilfeld BM. Relative Effects of Various Factors on Ice Ball Formation and Ablation Zone Size During Ultrasound-Guided Percutaneous Cryoneurolysis: A Laboratory Investigation to Inform Clinical Practice and Future Research. Pain Ther. 2023 Jun;12(3):771-783. doi: 10.1007/s40122-023-00497-y. Epub 2023 Mar 31. PMID 37000371
- [Derived] Ilfeld BM, Finneran JJ, Abdullah B, Vadakkan S, Alkabalan RA, Gabriel RA. Cryoanalgesia to treat phantom limb pain following a trans-femoral (above-knee) amputation: a randomized, sham-controlled pilot study. Reg Anesth Pain Med. 2025 Oct 13:rapm-2025-107116. doi: 10.1136/rapm-2025-107116. Online ahead of print. PMID 41033797